CLINICAL TRIAL: NCT00006180
Title: The P.O.W.E.R. STUDY (Premenopause, Osteopenia/Osteoporosis, Women, Alendronate, Depression)
Brief Title: Bone Loss in Premenopausal Women With Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 000203; 00-M-0203
Record Dates: First submitted 2000-08-17; First posted 2000-08-18 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-01-19

CONDITIONS: Depression; Healthy; Osteopenia; Osteoporosis
Keywords: Preventive Medicine; Women's Health; Bone Formation; Mood Disorders; Bone Resorption; Major Depression; Osteopenia; Osteoporosis; Bone Fracture; Bisphosphonate; Depression; Bone Density; Healthy Volunteer; HV; Normal Control
MeSH Terms: conditions — Depression; Bone Diseases, Metabolic; Osteoporosis; Mood Disorders; Bone Resorption; Depressive Disorder, Major; Fractures, Bone | interventions — Alendronate

INTERVENTIONS:
Drug: Alendronate

SUMMARY:
The purpose of this study is to determine whether women with major depression lose bone mass at a faster rate than women without depression. This study will also determine if the drug alendronate can maintain or increase bone mass in premenopausal women with major depression and osteoporosis.

Depression may be a major risk factor for osteoporosis; it is associated with abnormally elevated stress hormone levels that may contribute to bone loss. This study will evaluate bone mass in women with depression and healthy volunteers.

Participants will undergo psychiatric, medical, dietary, and stress hormone evaluations and bone mineral density (BMD) measurements.

Participants with depression will be divided into two groups: those with normal BMD and those with low BMD. Depressed participants with normal BMD will be compared to a control group of healthy premenopausal women with normal BMD and followed for 36 months. Dual energy X-ray absorptiometry (DEXA) determinations will be made at months 6, 12, 24 and 36; bone turnover and endocrine parameters of depression will be

measured every 3 to 6 months.

Participants with depression and low BMD will be randomly assigned to receive either alendronate or placebo (an inactive pill) once a week for 24 months. Participants will receive calcium and vitamin D supplements daily. DEXA determinations will be performed at screening, and at Months 6, 12, 18 and 24; bone turnover and endocrine parameters of depression will be measured every 3 to 6 months.

For both groups, up to four of the visits may optimally be done as inpatient stays of two nights. All remaining visits are as outpatients.

DETAILED DESCRIPTION:
This is a five-year study on the natural history of bone turn-over in depressed premenopausal women, ages 21 to 45 years, with normal bone mass, and the response to treatment with alendronate in depressed premenopausal women, ages 21 to 45 with low bone mass (as indicated by a bone mineral density (BMD) of negative 1.5 SD below peak bone mass at the spine and/or hip). Osteopenia is defined as a BMD at the spine and/or hip that is between negative 1.5 and negative 2.5 SD; osteoporosis is defined as a BMD that is below negative 2.5 SD at the spine and/or hip. During the initial screening, the women are evaluated for depression. Women who meet DSM-IV diagnostic criteria for Major Depressive Disorder as indicated by a structured psychiatric interview (SCID-IV and HAM-D), will then undergo a DEXA scan to determine BMD. Participants will be divided into four subcategories based on BMD results. Premenopausal depressed women with normal BMD (less than negative 1 SD below the average peak bone mass at the spine and/or hip) (Group B) will be matched by age, race, and body mass index to a control group of healthy, premenopausal, non-depressed women with normal bone mass (Group A). Groups A and B will be followed for 12 months with DEXA determinations every 6 months, measurements of bone turnover markers every 3 months, measurements of relevant endocrine parameters every 3 months, an exercise substudy at 0, 6, and 12 months, and collection of a DNA sample at one of the above visits.

Women with depression and low BMD (negative 1.5 SD below peak bone mass at the spine and/or hip) will enter a 12-month, placebo-controlled, clinical trial where they will be randomized either to blind alendronate 70 mg once a week (Group C) or blind placebo once a week (Group D). In addition to alendronate 70 mg once a week or placebo once a week, women in Groups C and D will also receive daily 500 mg of elemental calcium and 400 IU of vitamin D. DEXA determinations will be performed at Screening, Month 0, Month 6, and Month 12. Determination of biochemical markers of bone turnover and endocrine parameters relevant to depression will be performed at 0, 3, 6, 9 and 12 months. An exercise substudy will be performed at 0, 6, and 12 months. The collection of a DNA sample will also be performed at one of the above visits.

ELIGIBILITY:
* INCLUSION CRITERIA - DEPRESSED WOMEN:

The patient is a woman 21 to 45 years old on the date of the initial screening.

The patient is not postmenopausal.

She must be willing to practice an acceptable method of birth control, as appropriate (IUD, oral contraceptives, diaphragm, condoms, hormonal implants/injection, with the exception of subdermal levonorgestrel, sterilization) and have a negative serum pregnancy test at screening.

Women currently on estrogen/progestin contraceptive therapy must have been on a stable regimen of estrogen/progestin for at least 6 months prior to enter the study.

The patient understands the procedures and the risks of the study and has been informed that, alternatively, she may freely elect to be treated with the currently available treatments by her physician.

The patient voluntarily agrees to participate in the study.

INCLUSION CRITERIA RELATED TO THE PSYCHIATRIC STATUS:

The patient had at least one episode of major depression within the last 3 years (DSM-IV). In addition, the subject has a past history (prior to the last 3 years) of at least one major depressive episode lasting more than 2 weeks.

With the exception of depression, the patient is in good health, based on medical history, physical examination, and laboratory screening evaluation.

The patient has a physician; either a family doctor, a psychiatrist, a psychotherapist, or another qualified health care professional who can provide medical treatment for depression. If the subject is not receiving any medical care for depression, a member of the NIH team will help the patient identify one and will work closely with this professional during the study.

The patient can be on pharmacological antidepressant therapy, as medically indicated and prescribed by her primary physician or health professional. It is not a requirement of this study for subjects to stop antidepressant treatment, unless it is medically indicated for reasons such as the medication is ineffective, not well tolerated, or the patient no longer needs such treatment. This decision will be based upon their physician's evaluation.

Patients starting a new antidepressant medication(s) should be on this treatment for 4-6 weeks prior to enrollment.

Carbamazepine, valproic acid or thyroid hormones used as adjunctive therapy for treatment of depression are allowed.

Women with a current or recent (within the past 3 years) history of alcohol or drug abuse are eligible if, in the opinion of the principal investigator, this condition is not likely to impair patient compliance or if the participation in the study does not pose additional risks to the subject.

INCLUSION CRITERIA RELATED TO THE BONE STATUS:

The patient has spinal anatomy suitable for dual-energy x-ray absorptiometry (DEXA) densitometry of the lumbar spine, with no evidence of vertebral fractures in at least three vertebrae. Significant scoliosis, bony trauma, osteoarthritis, and sequelae of orthopedic procedures that result in anatomy unsuitable for accurate bone densitometry, must be absent from the lumbar spine.

The patient has osteopenia or osteoporosis, as indicated by a bone mineral density at the spine that is between 1.5 and 5 standard deviations below peak bone mass, or history of an osteoporotic vertebral or hip fracture. Patients whose eligibility is based only on a prevalent vertebral fracture will have the fracture confirmed by a radiologist.

EXCLUSION CRITERIA - DEPRESSED WOMEN:

GENERAL EXCLUSION CRITERIA:

The patient is, in the opinion of the investigator, mentally or legally incapacitated such that informed consent cannot be obtained.

Pregnancy or breast-feeding.

Menopause.

The patient plans to move within the next 12 months to a location which could impair a continued follow-up.

The patient has a history of or evidence for an illness or has significant abnormalities on prestudy clinical or laboratory evaluations, which, in the opinion of the principal investigator, might complicate the interpretation of the data or pose additional risk to the subject.

The patient has any of the following medical conditions: any malabsorption syndrome, significant genitourinary, renal (serum creatinine greater than or equal to 1.6 mg/dL), hepatic, or pulmonary disease; uncontrolled hypertension; uncontrolled diabetes mellitus; decompensated heart failure; clinically significant arrhythmias; unstable angina, any immunodeficiency syndrome including AIDS.

The patient has received any drug of investigation within 30 days of the start of the study.

The use of subdermal levonorgestrel and similar preparations.

EXCLUSION CRITERIA RELATED TO THE PSYCHIATRIC STATUS:

The patient does not have an outside care provider for treatment of depression.

The patient is judged to be at suicidal risk, as clinically evident or indicated by a score of 4 at the Hamilton Scale, question 3 (suicide), or by reports of suicidal intent during SCID-IV interview.

The patient has a history suggesting potential for self-harm or violence towards others.

The patient currently has psychotic depression (e.g. hallucinations, delusions).

The patient has schizoaffective disorder.

Patients with a diagnosis of active anorexia nervosa, bulimia or any other eating disorder are not eligible.

Patients with a diagnosis of bipolar disorders type 1 or type 2 or any psychotic disorder other than psychotic depression are not eligible.

Women with a current or recent (within the past 3 years) history of alcohol or drug dependence are not eligible.

EXCLUSION CRITERIA RELATED TO THE BONE STATUS OR THE USE OF ALENDRONATE:

The patient is affected by severe osteoporosis, as indicated by a history of recurrent non-traumatic fractures and/or a BMD value which is below 4 SD the peak bone mass at the spine and/or the hip.

The patient has a history of recent major upper gastrointestinal (GI) (esophagus, stomach, duodenum) mucosal erosive disease. As defined by (1) significant upper GI bleeding within the last year resulting in hospitalization and/or transfusion. (2) Recurrent ulcer disease documented by radiographic or endoscopic means (two episodes in the last two years, or any documented ulcer in the preceeding 3 months). (3) Uncontrolled dyspepsia currently treated on a daily basis. (4) Esophageal or gastric variceal disease or (5) esophageal stricture, achalasia, or severe esophageal motor dysfunction. (This only applies to Group C and D)

The patient has a history of cancer with the following exceptions: (1) superficial basal or squamous cell carcinoma of the skin that was treated, and (2) other malignancies treated at least 10 years ago without any evidence of recurrence.

The patient has a history of, or evidence for, metabolic bone disease (other than low bone mineral density) including, but not limited to uncontrolled hyper- or hypocalcemia, hyper- or hypoparathyroidism, Paget's disease of bone, osteomalacia, or osteogenesis imperfecta. Patients with surgically cured hyperparathyrodism due to parathyroid adenoma (at least one year prior to randomization) are eligible for inclusion in the trial. Patients with well-controlled hyper- or hypothyrodism, as indicated by clinical evaluation and normal plasma TSH level are eligible for inclusion in the trial.

The patient has received treatment prior to enrollment in the study that might have influenced bone turnover including:

Beginning a regimen (for more than 2 consecutive weeks) within the last 6 months, of any estrogen preparation including mixed estrogen agonist/antagonist, (e.g., tamoxifen or raloxifene) or progestins.

Having used within the last 6 months any of the following: anabolic steroids (including DHEA and other weaker analogs), calcitonin, calcitriol, alfacalcidol, excess vitamin A (greater than 10,000 units/day) or vitamin D (greater than 1,000 units/day), cyclosporine, or anticonvulsivants.

The patient is on a thyroid hormone for treatment of a thyroid condition, unless the patient has received a stable dose for the last 6 weeks prior to study enrollment, and is euthyroid, as documented by an ultrasensitive TSH serum assay.

The patient is on fluoride at a dose greater than 1 mg/day any time (fluoride taken greater than 3 months ago for less than 1 week is acceptable).

The patient has a history of glucocorticoid treatment for more than 1 month, within 6 months prior to study start (patients who received therapeutic glucocorticoids in the past must be considered unlikely to need glucocorticoid treatment during the course of the study).

Any previous treatment with bisphophonates for more than 2 weeks.

The patient's screening 25-hydroxyvitamin D level is less than 15 ng/mL unless 24-h urine calcium and serum PTH, calcium, and alkaline phosphatase are all within the normal range.

The patient is not able to stand or sit upright for at least 30 minutes.

The patient has a body weight greater than 137 kg, due to limitations in the accuracy of DEXA measurements above this body weight.

EXCLUSION CRITERIA RELATED TO THE EXERCISE (COOPER) TEST:

Subjects on beta-blockers will not be eligible to participate in the 12-min test.

INCLUSION CRITERIA - HEALTHY CONTROL WOMEN:

Healthy control women must be of good physical health; specifically, no history of any DSM-IV diagnoses, including but not limited to depression and anorexia nervosa.

They also must have normal bone density, no history of osteoporotic fractures, and be willing to be on a valid contraceptive method.

EXCLUSION CRITERIA - HEALTHY CONTROL WOMEN:

Control women should not have any of the risk factors for bone loss such as smoking, alcohol abuse, dietary imbalances unless the risk factor is present only to a mild extent.

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 220
Dates: Start 2000-08-10; Study Completion 2007-01-19

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Chrousos GP, Gold PW. The concepts of stress and stress system disorders. Overview of physical and behavioral homeostasis. JAMA. 1992 Mar 4;267(9):1244-52. PMID 1538563
- [Derived] Cizza G, Mistry S, Nguyen VT, Eskandari F, Martinez P, Torvik S, Reynolds JC, Gold PW, Sinaii N, Csako G; POWER Study Group. Do premenopausal women with major depression have low bone mineral density? A 36-month prospective study. PLoS One. 2012;7(7):e40894. doi: 10.1371/journal.pone.0040894. Epub 2012 Jul 27. PMID 22848407
- [Derived] Cizza G, Ronsaville DS, Kleitz H, Eskandari F, Mistry S, Torvik S, Sonbolian N, Reynolds JC, Blackman MR, Gold PW, Martinez PE; P.O.W.E.R. (Premenopausal, Osteopenia/Osteoporosis, Women, Alendronate, Depression) Study Group. Clinical subtypes of depression are associated with specific metabolic parameters and circadian endocrine profiles in women: the power study. PLoS One. 2012;7(1):e28912. doi: 10.1371/journal.pone.0028912. Epub 2012 Jan 3. PMID 22235252
- [Derived] Eskandari F, Martinez PE, Torvik S, Phillips TM, Sternberg EM, Mistry S, Ronsaville D, Wesley R, Toomey C, Sebring NG, Reynolds JC, Blackman MR, Calis KA, Gold PW, Cizza G; Premenopausal, Osteoporosis Women, Alendronate, Depression (POWER) Study Group. Low bone mass in premenopausal women with depression. Arch Intern Med. 2007 Nov 26;167(21):2329-36. doi: 10.1001/archinte.167.21.2329. PMID 18039992